CLINICAL TRIAL: NCT00880191
Title: Phase III Double-Blind, Placebo-Controlled Study of Gabapentin for the Prevention of Delayed CINV (Chemotherapy Induced Nausea and Vomiting) in Patients Receiving Highly Emetogenic Chemotherapy
Brief Title: Gabapentin in Preventing Nausea and Vomiting in Patients Receiving Chemotherapy
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Alliance for Clinical Trials in Oncology (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: NCCTG-N08C3; NCI-2009-01110 (Registry Identifier: CTRP (Clinical Trials Reporting System)); CDR0000634077 (Registry Identifier: PDQ (Physician Data Query))
Record Dates: First submitted 2009-04-10; First posted 2009-04-13 (Estimated); Results first posted 2015-05-21 (Estimated); Last update posted 2016-07-06 (Estimated); Status verified 2016-07

CONDITIONS: Nausea and Vomiting; Unspecified Adult Solid Tumor, Protocol Specific
Keywords: nausea and vomiting; unspecified adult solid tumor, protocol specific
MeSH Terms: conditions — Nausea; Vomiting | interventions — Dexamethasone; Gabapentin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Arm I (Experimental): Patients receive oral dexamethasone with 5HT3 receptor antagonist and oral gabapentin once daily on day 1 of chemotherapy. Patients then receive oral dexamethasone twice daily with or without 5HT3 receptor antagonist on days 2-4, and oral gabapentin either two or three times daily on days 2-5 of chemotherapy.
  Interventions: Drug: dexamethasone; Drug: gabapentin
- Arm II (Experimental): Patients receive oral dexamethasone with 5HT3 receptor antagonist and oral placebo once daily on day 1 of chemotherapy. Patients then receive oral dexamethasone twice daily with or without 5HT3 receptor antagonist on days 2-4, and oral placebo either two or three times daily on days 2-5 of chemotherapy.
  Interventions: Drug: dexamethasone; Other: placebo

INTERVENTIONS:
Drug: dexamethasone — Given orally
Drug: gabapentin — Given orally
  Arms: Arm I
Other: placebo — Given orally
  Arms: Arm II

SUMMARY:
RATIONALE: Gabapentin may prevent or reduce delayed nausea and vomiting caused by chemotherapy. It is not yet known whether gabapentin is more effective than a placebo in preventing nausea and vomiting.

PURPOSE: This randomized phase III trial is studying the side effects of gabapentin and to see how well it works compared with a placebo in preventing nausea and vomiting in patients receiving chemotherapy.

DETAILED DESCRIPTION:
OBJECTIVES:

* To evaluate the effectiveness of gabapentin in controlling delayed chemotherapy-induced nausea and vomiting (CINV) in patients receiving highly emetogenic chemotherapy as defined by the percentage of complete responders (no emetic episodes and no rescue medication) on days 2 through 6 (five days after receipt of highly emetogenic chemotherapy) compared to an effective prophylactic regimen.
* To evaluate the effectiveness of gabapentin in controlling delayed CINV in patients receiving highly emetogenic chemotherapy as defined by the percentage of complete responders (no emetic episodes, no more than mild nausea, and no rescue medication) on days 2 through 6 compared to an effective prophylactic regimen.
* To compare the effectiveness of these regimens in controlling acute CINV on day 1 of treatment in these patients.
* To compare the use of rescue agents in these patients.
* To determine the tolerability of gabapentin in these patients.
* To evaluate the effect of gabapentin for delayed chemotherapy-induced nausea and vomiting on symptom distress and functional abilities in these patients.
* To compare alternative endpoints and methods for assessing nausea and vomiting and to determine how these measures compare to patient's satisfaction with symptom control, distress and function.

OUTLINE: This is a multicenter study. Patients are stratified according to gender, age (< 50 years vs > 50 years), history of alcoholism (yes vs no), and history of motion sickness or history of pregnancy induced nausea/vomiting (yes vs no). Patients are randomized to 1 of 2 treatment arms.

* Arm I: Patients receive oral dexamethasone with 5HT3 receptor antagonist and oral gabapentin once daily on day 1 of chemotherapy. Patients then receive oral dexamethasone twice daily with or without 5HT3 receptor antagonist on days 2-4, and oral gabapentin either two or three times daily on days 2-5 of chemotherapy.
* Arm II: Patients receive oral dexamethasone with 5HT3 receptor antagonist and oral placebo once daily on day 1 of chemotherapy. Patients then receive oral dexamethasone twice daily with or without 5HT3 receptor antagonist on days 2-4, and oral placebo either two or three times daily on days 2-5 of chemotherapy.

Patients complete a Functional Living Index - Emesis questionnaire, an overall satisfaction survey, and a side effect experience diary at baseline and on day 6. Patients also complete a nausea and vomiting diary at baseline and periodically during study therapy.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Scheduled to receive highly emetogenic chemotherapy

  * May be scheduled to receive prophylactic treatment for acute nausea and vomiting with a 5HT3 antagonist and dexamethasone 20 mg on day 1 of chemotherapy treatment
  * May be scheduled to receive multiple day chemotherapy regimens as long as the chemotherapy drugs given on the subsequent days have mild or no emetogenic potential
* Chemotherapy schedules must allow at least 7 days rest between courses involving administration of highly emetogenic chemotherapy
* No primary CNS malignancy and/or CNS metastasis

PATIENT CHARACTERISTICS:

* Eastern Cooperative Oncology Group (ECOG) performance status 0-2
* Life expectancy ≥ 3 months
* Creatinine ≤ 1.5 times upper limit of normal within the past 30 days
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* Ability to complete questionnaire(s) by his/herself or with assistance
* Able to swallow pills
* No epilepsy or seizure history
* No gastrointestinal obstruction, active peptic ulcer disease, or uncontrolled heartburn
* No history of nausea and/or vomiting related to any kind of chemotherapy
* No nausea or vomiting within the past 3 days
* No history of allergic or other adverse reaction to gabapentin or pregabalin

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics
* No prior moderate or highly emetogenic chemotherapy
* No prior or concurrent aprepitant or any other NK-1 receptor antagonist
* At least 1 months since prior and no concurrent gabapentin, pregabalin, or other anticonvulsants
* At least 7 days since prior and no concurrent pelvic or abdominal radiotherapy
* At least 3 days since prior antiemetics
* No concurrent or planned use of lorazepam, diphenhydramine, eszopiclone, and/or dronabinol during the 6 days of this study, except for treatment of breakthrough nausea and vomiting

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 430 (Actual)
Dates: Start 2009-04; Primary Completion 2011-03 (Actual); Study Completion 2015-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Debra Barton, RN, PhD, AOCN, FAAN, Study Chair — Mayo Clinic
Locations (247):
- United States (247):
  - Mayo Clinic Scottsdale, Scottsdale, Arizona
  - Aurora Presbyterian Hospital, Aurora, Colorado
  - Boulder Community Hospital, Boulder, Colorado
  - Penrose Cancer Center at Penrose Hospital, Colorado Springs, Colorado
  - St. Anthony Central Hospital, Denver, Colorado
  - Porter Adventist Hospital, Denver, Colorado
  - Presbyterian - St. Luke's Medical Center, Denver, Colorado
  - St. Joseph Hospital, Denver, Colorado
  - Rose Medical Center, Denver, Colorado
  - CCOP - Colorado Cancer Research Program, Denver, Colorado
  - Swedish Medical Center, Englewood, Colorado
  - Poudre Valley Hospital, Fort Collins, Colorado
  - Front Range Cancer Specialists, Fort Collins, Colorado
  - St. Mary's Regional Cancer Center at St. Mary's Hospital and Medical Center, Grand Junction, Colorado
  - North Colorado Medical Center, Greeley, Colorado
  - Sky Ridge Medical Center, Lone Tree, Colorado
  - Hope Cancer Care Center at Longmont United Hospital, Longmont, Colorado
  - McKee Medical Center, Loveland, Colorado
  - St. Mary - Corwin Regional Medical Center, Pueblo, Colorado
  - North Suburban Medical Center, Thornton, Colorado
  - Exempla Lutheran Medical Center, Wheat Ridge, Colorado
  - Saint Francis/Mount Sinai Regional Cancer Center at Saint Francis Hospital and Medical Center, Hartford, Connecticut
  - Mayo Clinic - Jacksonville, Jacksonville, Florida
  - MBCCOP - Medical College of Georgia Cancer Center, Augusta, Georgia
  - Rush-Copley Cancer Care Center, Aurora, Illinois
  - Illinois CancerCare - Bloomington, Bloomington, Illinois
  - St. Joseph Medical Center, Bloomington, Illinois
  - Graham Hospital, Canton, Illinois
  - Illinois CancerCare - Canton, Canton, Illinois
  - Illinois CancerCare - Carthage, Carthage, Illinois
  - Memorial Hospital, Carthage, Illinois
  - Eureka Community Hospital, Eureka, Illinois
  - Illinois CancerCare - Eureka, Eureka, Illinois
  - Galesburg Clinic, PC, Galesburg, Illinois
  - Illinois CancerCare - Galesburg, Galesburg, Illinois
  - Illinois CancerCare - Havana, Havana, Illinois
  - Mason District Hospital, Havana, Illinois
  - Illinois CancerCare - Kewanee Clinic, Kewanee, Illinois
  - Illinois CancerCare - Macomb, Macomb, Illinois
  - McDonough District Hospital, Macomb, Illinois
  - Trinity Cancer Center at Trinity Medical Center - 7th Street Campus, Moline, Illinois
  - Moline, Illinois
  - Illinois CancerCare - Monmouth, Monmouth, Illinois
  - BroMenn Regional Medical Center, Normal, Illinois
  - Community Cancer Center, Normal, Illinois
  - Illinois CancerCare - Community Cancer Center, Normal, Illinois
  - Community Hospital of Ottawa, Ottawa, Illinois
  - Oncology Hematology Associates of Central Illinois, PC - Ottawa, Ottawa, Illinois
  - Cancer Treatment Center at Pekin Hospital, Pekin, Illinois
  - Illinois CancerCare - Pekin, Pekin, Illinois
  - Proctor Hospital, Peoria, Illinois
  - CCOP - Illinois Oncology Research Association, Peoria, Illinois
  - Oncology Hematology Associates of Central Illinois, PC - Peoria, Peoria, Illinois
  - Methodist Medical Center of Illinois, Peoria, Illinois
  - OSF St. Francis Medical Center, Peoria, Illinois
  - Illinois CancerCare - Peru, Peru, Illinois
  - Illinois Valley Community Hospital, Peru, Illinois
  - Illinois CancerCare - Princeton, Princeton, Illinois
  - Perry Memorial Hospital, Princeton, Illinois
  - Illinois CancerCare - Spring Valley, Spring Valley, Illinois
  - CCOP - Carle Cancer Center, Urbana, Illinois
  - St. Francis Hospital and Health Centers - Beech Grove Campus, Beech Grove, Indiana
  - Elkhart Clinic, LLC, Elkhart, Indiana
  - Michiana Hematology-Oncology, PC - Elkhart, Elkhart, Indiana
  - Elkhart General Hospital, Elkhart, Indiana
  - Howard Community Hospital, Kokomo, Indiana
  - Center for Cancer Therapy at LaPorte Hospital and Health Services, La Porte, Indiana
  - Saint Anthony Memorial Health Centers, Michigan City, Indiana
  - Michiana Hematology-Oncology, PC - South Bend, Mishawaka, Indiana
  - Saint Joseph Regional Medical Center, Mishawaka, Indiana
  - Michiana Hematology Oncology PC - Plymouth, Plymouth, Indiana
  - Reid Hospital & Health Care Services, Richmond, Indiana
  - CCOP - Northern Indiana CR Consortium, South Bend, Indiana
  - Memorial Hospital of South Bend, South Bend, Indiana
  - South Bend Clinic, South Bend, Indiana
  - Michiana Hematology Oncology PC - La Porte, Westville, Indiana
  - McFarland Clinic, PC, Ames, Iowa
  - Bettendorf, Iowa
  - Medical Oncology and Hematology Associates - West Des Moines, Clive, Iowa
  - CCOP - Iowa Oncology Research Association, Des Moines, Iowa
  - John Stoddard Cancer Center at Iowa Methodist Medical Center, Des Moines, Iowa
  - Medical Oncology and Hematology Associates at John Stoddard Cancer Center, Des Moines, Iowa
  - Medical Oncology and Hematology Associates at Mercy Cancer Center, Des Moines, Iowa
  - Mercy Cancer Center at Mercy Medical Center - Des Moines, Des Moines, Iowa
  - John Stoddard Cancer Center at Iowa Lutheran Hospital, Des Moines, Iowa
  - Siouxland Hematology-Oncology Associates, LLP, Sioux City, Iowa
  - Mercy Medical Center - Sioux City, Sioux City, Iowa
  - St. Luke's Regional Medical Center, Sioux City, Iowa
  - Cancer Center of Kansas, PA - Chanute, Chanute, Kansas
  - Cancer Center of Kansas, PA - Dodge City, Dodge City, Kansas
  - Cancer Center of Kansas, PA - El Dorado, El Dorado, Kansas
  - Cancer Center of Kansas - Fort Scott, Fort Scott, Kansas
  - Cancer Center of Kansas-Independence, Independence, Kansas
  - Cancer Center of Kansas, PA - Kingman, Kingman, Kansas
  - Lawrence Memorial Hospital, Lawrence, Kansas
  - Cancer Center of Kansas, PA - Liberal, Liberal, Kansas
  - Cancer Center of Kansas, PA - Newton, Newton, Kansas
  - Cancer Center of Kansas, PA - Parsons, Parsons, Kansas
  - Cancer Center of Kansas, PA - Pratt, Pratt, Kansas
  - Cancer Center of Kansas, PA - Salina, Salina, Kansas
  - Cancer Center of Kansas, PA - Wellington, Wellington, Kansas
  - Cancer Center of Kansas, PA - Medical Arts Tower, Wichita, Kansas
  - Cancer Center of Kansas, PA - Wichita, Wichita, Kansas
  - CCOP - Wichita, Wichita, Kansas
  - Via Christi Cancer Center at Via Christi Regional Medical Center, Wichita, Kansas
  - Cancer Center of Kansas, PA - Winfield, Winfield, Kansas
  - Hickman Cancer Center at Bixby Medical Center, Adrian, Michigan
  - Saint Joseph Mercy Cancer Center, Ann Arbor, Michigan
  - CCOP - Michigan Cancer Research Consortium, Ann Arbor, Michigan
  - Oakwood Cancer Center at Oakwood Hospital and Medical Center, Dearborn, Michigan
  - Green Bay Oncology, Limited - Escanaba, Escanaba, Michigan
  - Genesys Hurley Cancer Institute, Flint, Michigan
  - Hurley Medical Center, Flint, Michigan
  - Van Elslander Cancer Center at St. John Hospital and Medical Center, Grosse Pointe Woods, Michigan
  - Dickinson County Healthcare System, Iron Mountain, Michigan
  - Foote Memorial Hospital, Jackson, Michigan
  - Haematology-Oncology Associates of Ohio and Michigan, PC, Lambertville, Michigan
  - Sparrow Regional Cancer Center, Lansing, Michigan
  - St. Mary Mercy Hospital, Livonia, Michigan
  - Community Cancer Center of Monroe, Monroe, Michigan
  - Mercy Memorial Hospital - Monroe, Monroe, Michigan
  - Michiana Hematology Oncology PC - Niles, Niles, Michigan
  - St. Joseph Mercy Oakland, Pontiac, Michigan
  - Mercy Regional Cancer Center at Mercy Hospital, Port Huron, Michigan
  - Seton Cancer Institute at Saint Mary's - Saginaw, Saginaw, Michigan
  - Lakeland Regional Cancer Care Center - St. Joseph, Saint Joseph, Michigan
  - Lakeside Cancer Specialists, PLLC, Saint Joseph, Michigan
  - St. John Macomb Hospital, Warren, Michigan
  - Alexandria, Minnesota
  - MeritCare Bemidji, Bemidji, Minnesota
  - Fairview Ridges Hospital, Burnsville, Minnesota
  - Mercy and Unity Cancer Center at Mercy Hospital, Coon Rapids, Minnesota
  - Duluth Clinic Cancer Center - Duluth, Duluth, Minnesota
  - CCOP - Duluth, Duluth, Minnesota
  - Miller - Dwan Medical Center, Duluth, Minnesota
  - Fairview Southdale Hospital, Edina, Minnesota
  - Fergus Falls Medical Group, PA, Fergus Falls, Minnesota
  - Mercy and Unity Cancer Center at Unity Hospital, Fridley, Minnesota
  - Hutchinson Area Health Care, Hutchinson, Minnesota
  - Immanuel St. Joseph's, Mankato, Minnesota
  - HealthEast Cancer Care at St. John's Hospital, Maplewood, Minnesota
  - Minnesota Oncology Hematology, PA - Maplewood, Maplewood, Minnesota
  - Virginia Piper Cancer Institute at Abbott - Northwestern Hospital, Minneapolis, Minnesota
  - Hennepin County Medical Center - Minneapolis, Minneapolis, Minnesota
  - Hubert H. Humphrey Cancer Center at North Memorial Outpatient Center, Robbinsdale, Minnesota
  - Mayo Clinic Cancer Center, Rochester, Minnesota
  - CentraCare Clinic - River Campus, Saint Cloud, Minnesota
  - Coborn Cancer Center, Saint Cloud, Minnesota
  - CCOP - Metro-Minnesota, Saint Louis Park, Minnesota
  - Park Nicollet Cancer Center, Saint Louis Park, Minnesota
  - Regions Hospital Cancer Care Center, Saint Paul, Minnesota
  - United Hospital, Saint Paul, Minnesota
  - St. Francis Cancer Center at St. Francis Medical Center, Shakopee, Minnesota
  - Ridgeview Medical Center, Waconia, Minnesota
  - Willmar Cancer Center at Rice Memorial Hospital, Willmar, Minnesota
  - Minnesota Oncology Hematology, PA - Woodbury, Woodbury, Minnesota
  - Missouri Baptist Cancer Center, St Louis, Missouri
  - Arch Medical Services, Incorporated at Center for Cancer Care and Research, St Louis, Missouri
  - Comprehensive Cancer Care, PC, St Louis, Missouri
  - Cancer Resource Center - Lincoln, Lincoln, Nebraska
  - CCOP - Missouri Valley Cancer Consortium, Omaha, Nebraska
  - Immanuel Medical Center, Omaha, Nebraska
  - Alegant Health Cancer Center at Bergan Mercy Medical Center, Omaha, Nebraska
  - Creighton University Medical Center, Omaha, Nebraska
  - Lovelace Medical Center - Downtown, Albuquerque, New Mexico
  - University of New Mexico Cancer Center, Albuquerque, New Mexico
  - Rutherford Hospital, Rutherfordton, North Carolina
  - Bismarck Cancer Center, Bismarck, North Dakota
  - Medcenter One Hospital Cancer Care Center, Bismarck, North Dakota
  - Mid Dakota Clinic, PC, Bismarck, North Dakota
  - St. Alexius Medical Center Cancer Center, Bismarck, North Dakota
  - CCOP - MeritCare Hospital, Fargo, North Dakota
  - MeritCare Broadway, Fargo, North Dakota
  - Altru Cancer Center at Altru Hospital, Grand Forks, North Dakota
  - Mary Rutan Hospital, Bellefontaine, Ohio
  - Wood County Oncology Center, Bowling Green, Ohio
  - Adena Regional Medical Center, Chillicothe, Ohio
  - North Coast Cancer Care - Clyde, Clyde, Ohio
  - Riverside Methodist Hospital Cancer Care, Columbus, Ohio
  - CCOP - Columbus, Columbus, Ohio
  - Grant Medical Center Cancer Care, Columbus, Ohio
  - Mount Carmel Health - West Hospital, Columbus, Ohio
  - Doctors Hospital at Ohio Health, Columbus, Ohio
  - Grandview Hospital, Dayton, Ohio
  - Good Samaritan Hospital, Dayton, Ohio
  - David L. Rike Cancer Center at Miami Valley Hospital, Dayton, Ohio
  - Samaritan North Cancer Care Center, Dayton, Ohio
  - CCOP - Dayton, Dayton, Ohio
  - Grady Memorial Hospital, Delaware, Ohio
  - Community Cancer Center, Elyria, Ohio
  - Hematology Oncology Center, Elyria, Ohio
  - Blanchard Valley Medical Associates, Findlay, Ohio
  - Middletown Regional Hospital, Franklin, Ohio
  - Wayne Hospital, Greenville, Ohio
  - Charles F. Kettering Memorial Hospital, Kettering, Ohio
  - Fairfield Medical Center, Lancaster, Ohio
  - Lima Memorial Hospital, Lima, Ohio
  - Strecker Cancer Center at Marietta Memorial Hospital, Marietta, Ohio
  - Northwest Ohio Oncology Center, Maumee, Ohio
  - St. Luke's Hospital, Maumee, Ohio
  - Knox Community Hospital, Mount Vernon, Ohio
  - Licking Memorial Cancer Care Program at Licking Memorial Hospital, Newark, Ohio
  - Fisher-Titus Medical Center, Norwalk, Ohio
  - St. Charles Mercy Hospital, Oregon, Ohio
  - Toledo Clinic - Oregon, Oregon, Ohio
  - North Coast Cancer Care, Incorporated, Sandusky, Ohio
  - Community Hospital of Springfield and Clark County, Springfield, Ohio
  - Flower Hospital Cancer Center, Sylvania, Ohio
  - Mercy Hospital of Tiffin, Tiffin, Ohio
  - Toledo Hospital, Toledo, Ohio
  - St. Vincent Mercy Medical Center, Toledo, Ohio
  - Medical University of Ohio Cancer Center, Toledo, Ohio
  - CCOP - Toledo Community Hospital, Toledo, Ohio
  - St. Anne Mercy Hospital, Toledo, Ohio
  - Toledo Clinic, Incorporated - Main Clinic, Toledo, Ohio
  - UVMC Cancer Care Center at Upper Valley Medical Center, Troy, Ohio
  - Fulton County Health Center, Wauseon, Ohio
  - Mount Carmel St. Ann's Cancer Center, Westerville, Ohio
  - Clinton Memorial Hospital, Wilmington, Ohio
  - United States Air Force Medical Center - Wright-Patterson, Wright-Patterson AFB, Ohio
  - Ruth G. McMillan Cancer Center at Greene Memorial Hospital, Xenia, Ohio
  - Genesis - Good Samaritan Hospital, Zanesville, Ohio
  - Natalie Warren Bryant Cancer Center at St. Francis Hospital, Tulsa, Oklahoma
  - AnMed Cancer Center, Anderson, South Carolina
  - CCOP - Upstate Carolina, Spartanburg, South Carolina
  - Gibbs Regional Cancer Center at Spartanburg Regional Medical Center, Spartanburg, South Carolina
  - Medical X-Ray Center, PC, Sioux Falls, South Dakota
  - Sanford Cancer Center at Sanford USD Medical Center, Sioux Falls, South Dakota
  - Fredericksburg Oncology, Incorporated, Fredericksburg, Virginia
  - Virginia Commonwealth University Massey Cancer Center, Richmond, Virginia
  - Marshfield Clinic - Chippewa Center, Chippewa Falls, Wisconsin
  - Marshfield Clinic Cancer Care at Regional Cancer Center, Eau Claire, Wisconsin
  - Green Bay Oncology, Limited at St. Vincent Hospital Regional Cancer Center, Green Bay, Wisconsin
  - Green Bay Oncology, Limited at St. Mary's Hospital, Green Bay, Wisconsin
  - St. Mary's Hospital Medical Center - Green Bay, Green Bay, Wisconsin
  - St. Vincent Hospital Regional Cancer Center, Green Bay, Wisconsin
  - Holy Family Memorial Medical Center Cancer Care Center, Manitowoc, Wisconsin
  - Bay Area Cancer Care Center at Bay Area Medical Center, Marinette, Wisconsin
  - Marshfield Clinic - Marshfield Center, Marshfield, Wisconsin
  - Marshfield Clinic - Lakeland Center, Minocqua, Wisconsin
  - Green Bay Oncology, Limited - Oconto Falls, Oconto Falls, Wisconsin
  - Ministry Medical Group at Saint Mary's Hospital, Rhinelander, Wisconsin
  - Marshfield Clinic - Indianhead Center, Rice Lake, Wisconsin
  - Marshfield Clinic at Saint Michael's Hospital, Stevens Point, Wisconsin
  - Green Bay Oncology, Limited - Sturgeon Bay, Sturgeon Bay, Wisconsin
  - Marshfield Clinic - Weston Center, Weston, Wisconsin
  - Marshfield Clinic - Wisconsin Rapids Center, Wisconsin Rapids, Wisconsin

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 430 patients were enrolled on this study. There are 17 cancelled patients, 7 on the gabapentin arm and 10 on the placebo arm.
Groups:
- Gabapentin: Patients receive oral dexamethasone with 5HT3 receptor antagonist and oral gabapentin once daily on day 1 of chemotherapy. Patients then receive oral dexamethasone twice daily with or without 5HT3 receptor antagonist on days 2-4, and oral gabapentin either two or three times daily on days 2-5 of chemotherapy.
  > dexamethasone: Given orally
  > gabapentin: Given orally
- Placebo: Patients receive oral dexamethasone with 5HT3 receptor antagonist and oral placebo once daily on day 1 of chemotherapy. Patients then receive oral dexamethasone twice daily with or without 5HT3 receptor antagonist on days 2-4, and oral placebo either two or three times daily on days 2-5 of chemotherapy.
  > dexamethasone: Given orally
  > placebo: Given orally
Period: Overall Study
Arm/Group | Gabapentin | Placebo
Started | 207 | 206
Available for Primary Endpoint Analysis | 207 | 206
Completed | 194 | 198
Not Completed | 13 | 8
Not completed — Refused further treatment | 4 | 1
Not completed — Adverse Event | 8 | 6
Not completed — Hospitalization/efficacy | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Gabapentin: Patients receive oral dexamethasone with 5HT3 receptor antagonist and oral gabapentin once daily on day 1 of chemotherapy. Patients then receive oral dexamethasone twice daily with or without 5HT3 receptor antagonist on days 2-4, and oral gabapentin either two or three times daily on days 2-5 of chemotherapy.> dexamethasone: Given orally> gabapentin: Given orally
- Placebo: Patients receive oral dexamethasone with 5HT3 receptor antagonist and oral placebo once daily on day 1 of chemotherapy. Patients then receive oral dexamethasone twice daily with or without 5HT3 receptor antagonist on days 2-4, and oral placebo either two or three times daily on days 2-5 of chemotherapy.> dexamethasone: Given orally> placebo: Given orally
- Total: Total of all reporting groups
Arm/Group | Gabapentin | Placebo | Total
Number analyzed (Participants) | 207 | 206 | 413
Age, Customized [Number; unit: participants]
  <50 Years | 57 | 58 | 115
  >=50 Years | 150 | 148 | 298
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 145 | 145 | 290
  Male | 62 | 61 | 123
Region of Enrollment [Number; unit: participants]
  United States | 207 | 206 | 413

OUTCOME MEASURES:

1. Primary Outcome: Comparison of Percentage of Complete Responders
Description: Complete response being defined as no emetic episodes and no use of rescue therapy for days 2 through 6. If a patient does not complete the study or does not provide complete data, they will be assumed to be a non-responder.
Time Frame: Days 2 through 6
Measure: Number; unit: percentage of participants
Arm/Group | Gabapentin | Placebo
Number analyzed (Participants) | 207 | 206
percentage of participants
  Response Days 2-6: No | 53.1 | 59.2
  Response Days 2-6: Yes | 46.9 | 40.8
Statistical Analysis 1: Comparison: Gabapentin vs Placebo; Complete Responders by Arm - Days 2-6, the primary analysis utilizes Fisher's exact test to compare the percentage of complete responders in each group (dex/gabapentin vs. dex/placebo), with complete response being defined as no emetic episodes and no use of rescue therapy for days 2 through 6. If a patient does not complete the study or does not provide complete data, they will be assumed to be a non-responder; Test type: Superiority or Other; p = 0.2344, Fisher Exact

2. Secondary Outcome: Complete Response
Description: The primary analysis described above was repeated using a slightly different alternate definition of complete response: no emetic episodes, no more than a mean of 2.5 on the nausea numeric analogue scale (0 - 10 (As bad as it could be)), and no rescue agents.
Time Frame: Days 2-6
Measure: Number; unit: percentage of participants
Arm/Group | Gabapentin | Placebo
Number analyzed (Participants) | 207 | 206
percentage of participants
  Response Days 2-6: No | 56 | 60.7
  Response Days 2-6: Yes | 44 | 39.3
Statistical Analysis 1: Comparison: Gabapentin vs Placebo; The primary analysis described above was repeated using a slightly different alternate definition of complete response: no emetic episodes, no more than a mean of 2.5 on the nausea numeric analogue scale, and no rescue agents; Test type: Superiority or Other; p = 0.3694, Fisher Exact

3. Secondary Outcome: Comparison of Percentages of Complete Responders on Day 1, vs. Days 1 Through 6 vs. Days 2 Through 6.
Description: The percentages of complete responders on day 1, vs. days 1 through 6 vs. days 2 through 6 will be compared between arms. Complete response being defined as no emetic episodes and no use of rescue therapy. If a patient does not complete the study or does not provide complete data, they will be assumed to be a non-responder.
Time Frame: Days 1 through 6
Measure: Number; unit: percentage of participants
Arm/Group | Gabapentin | Placebo
Number analyzed (Participants) | 207 | 206
percentage of participants
  Response Day 1: No | 32.4 | 33.5
  Response Day 1: Yes | 67.6 | 66.5
  Response Day 1-6: No | 60.4 | 63.6
  Response Day 1-6: Yes | 39.6 | 36.4
  Response Day 2-6: No | 62.3 | 65
  Response Day 2-6: Yes | 37.7 | 35

4. Secondary Outcome: Comparison of the Percentage of Patients Experiencing Emetic Episodes and the Percentage Needing Rescue Agents
Description: The percentage of patients experiencing emetic episodes and the percentage needing rescue agents was compared between groups.
Time Frame: Days1 through 6
Measure: Number; unit: percentage of participants
Arm/Group | Gabapentin | Placebo
Number analyzed (Participants) | 207 | 206
percentage of participants
  Rescue Agent Status: No | 55 | 47
  Rescue Agent Status: Yes | 45 | 53
  Emetic Status: No | 70 | 70
  Emetic Status: Yes | 30 | 30

5. Secondary Outcome: Comparison of Sum of the Daily Distress Questions as Well as the Individual Daily Responses
Description: The sum of the daily distress questions as well as the individual daily responses from the Nausea and Vomiting Diary (NVD) on a 0-10 scale (Lower score is better) will be compared.
Time Frame: Days 1 through 6
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Gabapentin | Placebo
Number analyzed (Participants) | 207 | 206
units on a scale
  NVD Nausea Distress Day 1 | 1.1 (2.3) | 1.2 (2.2)
  NVD Nausea Distress Day 2 | 0.9 (1.9) | 1.1 (1.7)
  NVD Nausea Distress Day 3 | 0.9 (1.9) | 1.2 (2.2)
  NVD Nausea Distress Day 4 | 0.7 (1.6) | 1.1 (1.9)
  NVD Nausea Distress Day 5 | 0.9 (1.9) | 1.1 (1.8)
  NVD Nausea Distress Day 6 | 0.8 (1.8) | 0.9 (1.7)
  NVD Nausea Distress Sum Days 1-6 | 5.1 (8.0) | 6.4 (8.9)

6. Secondary Outcome: Level of Satisfaction for the Control of Nausea.
Description: Level of satisfaction for the control of nausea with the mean severity of nausea over the six days in the diary (on a 0 - 10 scale, higher the better) as well as the nausea subscale on the Functional Living Index - Emesis (FLIE) questionnaire ( 1-7 scale, lower the better)
Time Frame: Days 1 through 6
Population: 203 patients in Gabapentin arm and 201 patients in Placebo arm submitted the data for this endpoint.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Gabapentin | Placebo
Number analyzed (Participants) | 203 | 201
units on a scale
  Satisfaction Nausea Control (0-10 scale) | 8.3 (2.8) | 8.1 (2.9)
  FLIE Nausea Subscale Day 6 | 2.8 (1.0) | 2.9 (1.0)

7. Secondary Outcome: Comparison of Daily Complete Response Endpoints
Description: Daily complete response is defined as no emetic episodes and no use of rescue therapy.
Time Frame: Days 1 through 6
Measure: Number; unit: percentage of participants
Arm/Group | Gabapentin | Placebo
Number analyzed (Participants) | 207 | 206
percentage of participants
  Response Day 1: No | 32.4 | 33.5
  Response Day 1: Yes | 67.6 | 66.5
  Response Day 2: No | 26.6 | 36.4
  Response Day 2: Yes | 73.4 | 63.6
  Response Day 3: No | 22.2 | 34.5
  Response Day 3: Yes | 77.8 | 65.5
  Response Day 4: No | 19.3 | 30.1
  Response Day 4: Yes | 80.7 | 69.9
  Response Day 5: No | 32.9 | 34.0
  Response Day 5: Yes | 67.1 | 66.0
  Response Day 6: No | 28.0 | 31.6
  Response Day 6: Yes | 72.0 | 68.4

ADVERSE EVENTS:
Arm/Group | Gabapentin | Placebo
Serious Adverse Events (participants affected / at risk) | 0/207 | 0/206
Other Adverse Events (participants affected / at risk) | 95/207 | 96/206
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Gabapentin (N=207) | Placebo (N=206)
Febrile neutropenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 1 (1) | 0 (0)
Vision blurred (Eye disorders) | 1 (1) | 0 (0)
Constipation (Gastrointestinal disorders) | 2 (2) | 2 (2)
Diarrhea (Gastrointestinal disorders) | 3 (3) | 1 (1)
Dyspepsia (Gastrointestinal disorders) | 6 (6) | 3 (3)
Flatulence (Gastrointestinal disorders) | 0 (0) | 1 (1)
Mucositis oral (Gastrointestinal disorders) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 5 (5) | 1 (1)
Vomiting (Gastrointestinal disorders) | 3 (3) | 3 (3)
Edema limbs (General disorders) | 19 (19) | 18 (18)
Fatigue (General disorders) | 2 (2) | 1 (1)
Localized edema (General disorders) | 3 (3) | 9 (9)
Pain (General disorders) | 0 (0) | 1 (1)
Device related infection (Infections and infestations) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 0 (0) | 1 (1)
Skin infection (Infections and infestations) | 0 (0) | 1 (1)
Alanine aminotransferase increased (Investigations) | 1 (1) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 0 (0) | 1 (1)
Blood glucose increased (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Serum sodium decreased (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Muscle weakness lower limb (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Ataxia (Nervous system disorders) | 13 (13) | 23 (23)
Depressed level of consciousness (Nervous system disorders) | 16 (16) | 17 (17)
Dizziness (Nervous system disorders) | 57 (58) | 59 (59)
Headache (Nervous system disorders) | 5 (5) | 3 (3)
Ischemia cerebrovascular (Nervous system disorders) | 1 (1) | 0 (0)
Speech disorder (Nervous system disorders) | 1 (1) | 0 (0)
Syncope (Nervous system disorders) | 0 (0) | 1 (1)
Confusion (Psychiatric disorders) | 1 (1) | 0 (0)
Renal failure (Renal and urinary disorders) | 0 (0) | 1 (1)
Allergic rhinitis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Hiccough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Dry skin (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Hypertension (Vascular disorders) | 1 (1) | 0 (0)
Thrombosis (Vascular disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes